CLINICAL TRIAL: NCT00052897
Title: A Phase I/II Trial of SGN-00101 in the Treatment of High-Grade Anal Intraepithelial Neoplasia (AIN) in HIV-Positive Individuals
Brief Title: SGN-00101 in Preventing Anal Cancer in Patients With HIV Who Have Anal Neoplasia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2012-02507; AMC-035; CDR0000258786 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2004-04

CONDITIONS: Anal Cancer
Keywords: anal cancer
MeSH Terms: conditions — Anus Neoplasms

ARMS (1):
- Arm I (Experimental): Patients receive SGN-00101 subcutaneously once on weeks 0, 4, and 8. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Cohorts of 5-6 patients receive escalating doses of SGN-00101 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 1 of 6 patients experience dose-limiting toxicity.
  Interventions: Biological: HspE7

INTERVENTIONS:
Biological: HspE7

SUMMARY:
Phase I/II trial to study the effectiveness of SGN-00101 in preventing anal cancer in HIV-positive patients who have high-grade anal neoplasia. Chemoprevention therapy is the use of certain drugs to try to prevent the development of cancer. SGN-00101 may be effective in preventing anal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the safety and maximum tolerated dose of SGN-00101 in HIV-positive patients with high-grade anal squamous intraepithelial lesions.

II. Determine clinical response and histologic/cytologic regression in patients treated with this drug.

III. Determine immune response in patients treated with this drug. IV. Determine the effect of this drug on HIV viral load and CD4 level in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive SGN-00101 subcutaneously once on weeks 0, 4, and 8. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 5-6 patients receive escalating doses of SGN-00101 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 1 of 6 patients experience dose-limiting toxicity.

Patients are followed at 1, 4, and 10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed high-grade anal squamous intraepithelial lesions (HSIL) with residual HSIL of the anal canal or margin by high-resolution anoscopy

  * Declined routine surgery or not a candidate for surgical excision of HSIL
* Documented evidence of HIV infection by one of the following methods:

  * Serologic (ELISA or western blot)
  * Culture
  * Quantitative polymerase chain reaction or bDNA assays
* HIV RNA no greater than 500 copies/mL
* CD4 at least 200 x 10^6/L
* Must have received stable highly active antiviral therapy (HAART) for at least 4 weeks before study

  * HAART defined as 3 or more agents, including a protease inhibitor or nonnucleoside reverse transcriptase inhibitor that is approved or available through expanded access combination antiviral therapy
* No prior history of invasive anal or cervical cancer
* No concurrent untreated cervical HSIL

PATIENT CHARACTERISTICS:

Age

* 18 and over

Life expectancy

* At least 12 months

Hematopoietic

* Hemoglobin at least 10 g/dL
* Platelet count at least 75,000/mm^3
* Absolute neutrophil count at least 1,000/mm^3

Hepatic

* AST and ALT no greater than 3 times upper limit of normal (ULN)

Renal

* Creatinine no greater than 1.5 times ULN

Immunologic

* No prior severe allergic reactions (i.e., anaphylactic response) to drugs or any other allergen
* No history of collagen-vascular or autoimmune disorder requiring treatment within the past 5 years
* No other concurrent illness that compromises the immune system
* No active serious opportunistic infection

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 forms of effective contraception during and for 3 months after study
* No concurrent participation in a conception process (e.g., active attempt to become pregnant or impregnate, sperm donation, or in vitro fertilization)
* No other concurrent medical or psychiatric illness that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunostimulants (including interferon or interleukin-12)

Chemotherapy

* More than 1 year since prior chemotherapy for cancer

Endocrine therapy

* No concurrent steroids that compromise immune function

  * Concurrent topical corticosteroids allowed if dose determined not to suppress immune function

Radiotherapy

* More than 1 year since prior radiotherapy for cancer

Other

* More than 30 days since other prior investigational agents
* No concurrent medications that suppress immune function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2002-12; Primary Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Palefsky, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Comprehensive Cancer Center, San Francisco, California, United States